CLINICAL TRIAL: NCT06115018
Title: The Efficacy and Maintain Effect of Oropharyngeal Rehabilitation on Obstructive Sleep Apnea Patients After Palatal Surgery
Brief Title: The Efficacy and Maintain Effect of OPR on OSA Patients After Palatal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi-Ju, Lai (Other)
Responsible Party: Sponsor-Investigator, Yi-Ju, Lai, Institute of Physical Education, Health and Leisure Studies, College of Management, National Cheng Kung University, Tainan, Taiwan, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-112-052
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Oropharyngeal rehabilitation; Computed tomography; Tongue muscle strength; Maintain effect
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palatal surgery group (Active Comparator): In the palatal surgery group, the participants will receive palatal surgery.To evaluate the effect of treatments on the severity of OSA, tongue muscle strength and the space of the upper airway, the participants will receive polysomonogrphy test, tongue muscle strength test and computed tomography. The time of evaluation will include baseline, 3 and 6 months after treatment.
  Interventions: Procedure: Palatal surgery
- Oropharyngeal rehabilitation group (Active Comparator): In the oropharyngeal rehabilitation (OPR) group, the participants will receive 12-week OPR. The OPR for the OPR group included three 30-minute sessions of OPR per day, and the exercise would be performed 3-5 days per week for 3 months. The performance of the home exercise will also be recorded by the force-sensing resistor. In addition to home exercise sessions, there will also be twice-weekly clinical visits to adjust the contents of OPR program and monitor training progress. To evaluate the effect of treatments on the severity of OSA, tongue muscle strength and the space of the upper airway, the participants will receive polysomonogrphy test, tongue muscle strength test and computed tomography. The time of evaluation will include baseline, 3 and 6 months after treatment.
  Interventions: Behavioral: Oropharyngeal rehabilitation
- Palatal surgery combined OPR group (Experimental): In the palatal surgery combined OPR group, the participants will receive palatal surgery, then 12-week OPR. The program of OPR for this group is as the same of OPR group.
  Interventions: Combination Product: Palatal surgery combined oropharyngeal rehabilitation

INTERVENTIONS:
Procedure: Palatal surgery — Palate surgery has evolved from the ablative partial palate resections, which favored the removal of the soft tissue that obstructed the upper airway (UA), to more recent innovative reconstructive procedures that not only address the level of palatal obstruction, but the type of palatal or lateral pharyngeal wall collapse.
  Arms: Palatal surgery group
Behavioral: Oropharyngeal rehabilitation — Oropharyngeal rehabilitation (OPR) focus on the upper airway muscle including tongue muscle, palatal muscles and paryngeal muscles. The OPR for the treatment groups included three 30-minute sessions of OPR per day, and the exercise would be performed 3-5 days per week for 3 months. The performance of the home exercise will also be recorded by the force-sensing resistor. In addition to home exercise sessions, there will also be twice-weekly clinical visits to adjust the contents of OPR program and monitor training progress.
  Arms: Oropharyngeal rehabilitation group
Combination Product: Palatal surgery combined oropharyngeal rehabilitation — Participants will receive palatal surgery and post-surgery oropharyngeal rehabilitation (OPR). The palatal surgery and OPR describe as above.
  Arms: Palatal surgery combined OPR group

SUMMARY:
The goal of this clinical trial is to evaluate the maintain effect of palatal surgery and oropharyngeal rehabilitation (OPR) by using the severity of obstructive sleep apnea (OSA), tongue muscle strength and the space of the upper airway in patients with OSA.The main questions it aims to answer are:

1. Will the severity of OSA, tongue muscle strength and the space of upper airway improve more in the palatal surgery combined OPR group than the other two groups?
2. Will The maintain effect of tongue muscle strength and the space of upper airway be better in the palatal surgery combined OPR group? Participants will be divided into 3 groups including palatal surgery combined OPR group, palatal surgery group and OPR group by the doctor's advice and their willingness.The OPR for the treatment groups included three 30-minute sessions of OPR per day, and the exercise would be performed 3-5 days per week for 3 months.

DETAILED DESCRIPTION:
Background: The pathophysiology of obstructive sleep apnea (OSA) includes anatomical and non-anatomical factors. The patients who are suitable for sleep surgery may have the non-anatomical factors at the same time. Oropharyngeal rehabilitation (OPR) for the extrinsic and intrinsic muscles of the tongue might mitigate sleep apnea by preventing airway collapse and reducing the volume of the tongue base. In addition, previous studies also suggested that increasing the tension of the tongue extrinsic/intrinsic muscles may decrease the collapsibility of the upper airway and further prevent airway collapse during sleep. Although palatal surgery and OPR both can improve the severity of OSA, there is lack of literatures about the maintain effect of palatal surgery combined OPR. The aim of this study is to evaluate the maintain effect by using the severity of OSA, tongue muscle strength and the space of the upper airway. Our team have developed force sensing resistor to record the times and frequency of OPR at home from 2022. However, the investigators have to use SD card to record data in the present version. The investigators will optimize the force sensing resistor to upload data to Google Drive by using wifi. In this way, the investigators will know the daily training situation and give feedback to participants immediately by using LINE.

Methods：Seventy-five adult OSA patients will be recruited for this study. Participants will be divided into 3 groups including palatal surgery combined OPR group, palatal surgery group and OPR group by the doctor's advice and their willingness. In the palatal surgery combined OPR group, the participants will receive the palatal surgery and 3-month OPR. In the palatal surgery group and OPR group, the participants will receive palatal surgery or 3-month OPR, respectively. The OPR for the treatment groups included three 30-minute sessions of OPR per day, and the exercise would be performed 3-5 days per week for 3 months. The performance of the home exercise will also be recorded by the force-sensing resistor. In addition to home exercise sessions, there will also be twice-weekly clinical visits to adjust the contents of OPR program and monitor training progress. To evaluate the effect of treatments on the severity of OSA, tongue muscle strength and the space of the upper airway, the participants will receive polysomonogrphy test, tongue muscle strength test and computed tomography. The time of evaluation will include baseline, 3 and 6 months after treatment.

Expected outcomes：

1. The severity of OSA, tongue muscle strength and the space of upper airway will improve more in the palatal surgery combined OPR group than the other two groups.
2. The maintain effect of tongue muscle strength and the space of upper airway is better in the palatal surgery combined OPR group.

ELIGIBILITY:
Inclusion Criteria:

* mild to severe obstructive sleep apnea patients

Exclusion Criteria:

* Chronic rhinosinusitis with nasal polyps
* Adenoidal hypertrophy
* Bilateral tonsile hypertrophy
* Morbid Obesity
* Drug or alcohol abuse in one year
* Pregnancy
* Severe lung disease
* Heart disease with high risk of exercise
* Neuromuscular disease that can't follow the exercise program
* Central or mixed sleep apnea

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG) | Single night (8 hours)
  PSG will include electroencephalography, electrooculography, electromyography, thoracic and abdominal respiratory inductance plethysmography, body position sensor-modified lead II electrocardiography, oronasal thermistor, nasal cannula pressure transducer, finger pulse oximetry. The detail descriptions of each measurement are in secondary outcome measure.
  From the abouve measurements, OSA severity, defined using AHI, will be diagnosed by sleep medicine specialists in the ear, nose, and throat (ENT) department. AHI denotes the number of instances of apnea and hypopnea per hour during sleep. Apnea was defined as a >90% decrease in airflow and a >10-s cessation of airflow, and hypopnea was defined as a >30% decrease in airflow and >3% decrease in oxygen desaturation or microarousal. AHI of 5 to <15, 15 to <30, ≥30 denotes mild, moderate, and severe OSA, respectively.
CT | 10-20 minutes
  Each participant will maintain their tongues in the resting position, without swallowing, during CT. Pharyngeal airway volume, minimal cross-sectional areas, minimal distance between the lateral pharyngeal wall on both sides, and minimal distance between the anterior and posterior pharyngeal wall on the tip of the epiglottis will be measured. The detail description of each measurement are in secondary outcome measure. Experienced radiologists will perform image reconstruction and data analysis.
Tongue muscle strength | 10 minutes
  Tongue muscle strength will be evaluated on the IOPI system (model 2.2; Northwest, Carnation, WA, USA). The participants will sit in a relaxed position, with their heads parallel to the horizontal plane and their feet on the ground. The evaluation probe will comprise a balloon and plastic catheter. The participants will squeeze the balloon for 3 s at maximum pressure. The maximum pressure of protrusion, lateralization, elevation, and depression will be considered the highest of three measurements, expressed in kilopascals.
Questionnaires (including Epworth Sleepiness Scale, Pittsburgh Sleep Questionnaire Index, Snore Outcomes Survey etc.) | 10 minutes
  We will use ESS to evaluate daytime sleepiness. We will use PSQI to assess sleep quality and patterns. SOS consists of eight items related to the frequency, duration, severity, and consequences associated with sleep-disordered breathing and specifically snoring. Because of the effect of sleep-disordered breathing on partners, a separate Spouse/Bed Partner Survey (SBPS), comprising three Likert-type items, will also be used.

SECONDARY OUTCOMES:
Electroencephalography from Polysomnography (PSG) | Single night (8 hours)
  Electroencephalogram (EEG) is a test that measures electrical activity in the brain using small, metal discs (electrodes) attached to the scalp. It will be used to determine the sleeping stages of the participants.
Electrooculography from Polysomnography (PSG) | Single night (8 hours)
  Electrooculography (EOG) is a technique for measuring the corneo-retinal standing potential that exists between the front and the back of the human eye. It will be used to know the participants is in repeat eye movement stage or non-repeat eye movement stage.
Electromyography from Polysomnography (PSG) | Single night (8 hours)
  Electromyography (EMG) is a technique for evaluating and recording the electrical activity produced by skeletal muscles. EMG will be used to evaluate limb movement during sleep. Surface EMG will be used in PSG.
Thoracic and abdominal respiratory inductance plethysmography from Polysomnography (PSG) | Single night (8 hours)
  Thoracic and abdominal respiratory inductance plethysmography is a method of monitoring pulmonary ventilation by measuring the movement of the chest and abdominal wall. Phase relation between thorax and abdomen classifies apnea/hypopnea events into central, mixed, and obstructive types.
Body position sensor-modified lead II electrocardiography from Polysomnography (PSG) | Single night (8 hours)
  It will be used to monitor the particiapants is in supine position or sidelying position.
Nasal cannula pressure transducer from PSG | Single night (8 hours)
  It will be used to monitor airflow from nose and evaluate epoch of hypopnea. Airflow is in L/sec.
Oronasal thermistor from PSG | Single night (8 hours)
  It will be used to monitor temperature from mouth and evaluate epoch of apnea. Temperature is in degree of celsius.
Finger pulse oximetry from PSG | Single night (8 hours)
  It will be used to evaluate SpO2. SpO2 is in %.
Pharyngeal airway volume | 10-20 minutes
  Pharyngeal airway volume from the hard palate to the epiglottis will be measured. Volume in cm cubed.
Minimal cross-sectional areas | 10-20 minutes
  The minimal cross-sectional areas on the tip of the epiglottis will be measured. Areas in cm.
Minimal distance between the lateral pharyngeal wall on both sides, and minimal distance between the anterior and posterior pharyngeal wall | 10-20 minutes
  Minimal distance between the lateral pharyngeal wall on both sides, and minimal distance between the anterior and posterior pharyngeal wall on the tip of the epiglottis will be measured. Distance in cm.
Epworth Sleepiness Scale (ESS) | 5 minutes
  ESS consists of eight situations measured on a scale of 0-3, representing no, occasional, common, and frequent sleepiness, respectively. The scores for the eight situations are totaled. Total scores of 0 to 10 points represent normal results, whereas total scores of 11-24 points indicate high levels of daytime sleepiness.
Pittsburgh Sleep Questionnaire Index (PSQI) | 5 minutes
  It consists of nine items covering seven domains: subjective sleep quality, sleep latency, sleep duration, sleep disturbances, habitual sleep efficiency, sleep medication use, and daytime dysfunction. The participants' responses were based on the coditions in the month prior. The total scores range from 0 to 21 points, and a total score of >5 points indicates poor sleep.
Snore Outcomes Survey (SOS) | 5 minutes
  SOS consists of eight items related to the frequency, duration, severity, and consequences associated with sleep-disordered breathing and specifically snoring. Because of the effect of sleep-disordered breathing on partners, a separate Spouse/Bed Partner Survey (SBPS), comprising three Likert-type items, was also used. The scores on the SOS and SBPS were normalized to the range of 0 (worst) to 100 points (best).

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Lai, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Other co-author in our study havn't made their decision yet.